CLINICAL TRIAL: NCT01056666
Title: Evaluation de l'Impact Sur la qualité de Vie de l'Utilisation d'un système Collecteur Conveen( étuis pénien Conveen Optima Avec Poches de Recueil Conveen) Chez Des Hommes Souffrant d'Une Incontinence Urinaire modérée ou sévère, Comparativement à Leur Protection Absorbante Habituelle
Brief Title: Conveen Optima Urisheaths With Collecting Bags Versus Absorbents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FR002CC
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Last update posted 2011-09-19 (Estimated); Status verified 2007-04

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conveen optima urisheaths (Experimental)
  Interventions: Device: Conveen Optima is a urisheath to be used together with a collecting bag for urine
- absorbent protections (Placebo Comparator): The patient use their usual absorbent protection as comparator. All brands are allowed.
  Interventions: Device: absorbent protection

INTERVENTIONS:
Device: Conveen Optima is a urisheath to be used together with a collecting bag for urine — Conveen optima urisheath is intended to be used together with a collecting bag for urine and to be changed on a daily basis
  Arms: Conveen optima urisheaths
Device: absorbent protection — The patient use his usual absorbent protection (same brand), and change it when needed
  Arms: absorbent protections

SUMMARY:
The objective of this investigation is to asses with validated scales, the impact on the quality of life of men suffering of moderate to severe incontinence of the use of Conveen Optima urisheath in comparison with their usual absorbent protection.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18
* Out clinic patient
* Patient using absorbent protection for his urinary incontinence
* Moderate to severe urinary incontinence (1 hour pad test > 10g)
* All kind of stable urinary incontinence
* Patient able to apply himself the device
* Patient able to understand the questions
* Patient having given his informed consent
* Patient whose overall treatment for his urinary incontinence is not modified during the study

Exclusion Criteria:

* Patient having a retracted penis
* Patient having skin problem on the penis
* Patient using urisheaths
* Bedridden patient
* Institutionalized patient
* Patient with indwelling catheter or under intermittent catheterisation
* Patient with fecal incontinence leading to the use of absorbent protection
* Patient suffering of urinary tract infection

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2007-06; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Impact on quality of life | Days 0, 15, 30

SECONDARY OUTCOMES:
Efficacy (leakages) | days 13, 14, 15 and days 28, 29, 30

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Costa, Professor, Principal Investigator — Hôpital Caremeau Nimes. France